CLINICAL TRIAL: NCT05741216
Title: Evaluation of Comfort of Ocular Lubricants in Symptomatic Contact Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEJ475-E006
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- OTF Test 1 (Experimental): One application of ocular lubricant to each eye at night for 5 consecutive nights
  Interventions: Other: OTF Ocular Lubricant
- OTF Test 2 (Experimental): One application of ocular lubricant to each eye at night for 5 consecutive nights
  Interventions: Other: OTF Ocular Lubricant
- OTF Test 3 (Experimental): One application of ocular lubricant to each eye at night for 5 consecutive nights
  Interventions: Other: OTF Ocular Lubricant
- Ocular lubricant (Active Comparator): One drop of ocular lubricant applied to each eye at night for 5 consecutive nights
  Interventions: Other: Ocular Lubricant

INTERVENTIONS:
Other: OTF Ocular Lubricant — Ocular lubricant in 1 of 3 test formulations
  Arms: OTF Test 1; OTF Test 2; OTF Test 3
Other: Ocular Lubricant — Commercially available ocular lubricant
  Other Names: SYSTANE™ Gel; Genteal™ Gel
  Arms: Ocular lubricant

SUMMARY:
The purpose of this study is to evaluate the ocular comfort of 3 ocular lubricants and a comparator.

DETAILED DESCRIPTION:
The expected duration of subject participation is at least 7 days. This study will be conducted in Australia and Canada.

ELIGIBILITY:
Key Inclusion Criteria:

* Is able to understand and sign an approved information consent letter;
* Habitually wears daily disposable soft contact lenses in both eyes
* Uses rewetting drops on a regular basis;
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Routinely sleeps in habitual contact lenses;
* Has any known active ocular disease and/or infection;
* Is pregnant or lactating;
* Other protocol specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
Ocular comfort | Up to Day 5
  Comfort will be rated using a visual analog scale (0-100) from 0-100, where 0=poor and 100=excellent.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Dry Eye, Study Director — Alcon Research, LLC
Locations (3):
- Australia (2):
  - School of Optometry and Vision, Sydney, New South Wales
  - Deakin Collaborative Eye Care Clinic, Deakin University, Waurn Ponds, Victoria
- School of Optometry and Vision Science, University of Waterloo, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No